CLINICAL TRIAL: NCT07349082
Title: Comparison of Sensory Block Onset Time Between Epidural and Dural Puncture Epidural (DPE) Anesthesia for Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Sensory Block Onset: Epidural vs Dural Puncture Epidural in Cesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Naufal Anasy, Principal Investigator, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NaufalRCT1
Record Dates: First submitted 2025-12-23; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cesarean Section
Keywords: cesarean section; epidural anesthesia; dural puncture epidural; sensory block onset; hemodynamic stability
MeSH Terms: interventions — Anesthesia; Anesthesia, Epidural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dural Puncture Epidural (DPE) Anesthesia (Experimental): Participants receive a dural puncture epidural (DPE) anesthesia for elective cesarean delivery.
  Interventions: Procedure: Dural Puncture Epidural (DPE) Anesthesia
- Epidural Anesthesia (Active Comparator): Participants receive a conventional epidural anesthesia for elective cesarean delivery.
  Interventions: Procedure: epidural anesthesia

INTERVENTIONS:
Procedure: Dural Puncture Epidural (DPE) Anesthesia — Dural puncture epidural (DPE) is a combined neuraxial technique that integrates spinal and epidural approaches to enhance the quality of sensory and motor blockade. The procedure begins with dural puncture using a 26-gauge Spinocan spinal needle at the L3-L4 lumbar interspace until cerebrospinal fluid (CSF) is observed, indicating a micro-dural lesion, after which the spinal needle is withdrawn. Subsequently, an epidural catheter is inserted using an 18-gauge Tuohy needle with the loss-of-resistance (LOR) technique using saline, and advanced 4-5 cm into the epidural space. The anesthetic agents administered are the same as those used in conventional epidural anesthesia. This DPE technique is operationalized to accelerate sensory block onset, improve motor block quality, and minimize complications compared with conventional epidural anesthesia.
  Arms: Dural Puncture Epidural (DPE) Anesthesia
Procedure: epidural anesthesia — Conventional epidural technique for elective cesarean delivery. Epidural anesthesia is a neuraxial technique used for analgesia or anesthesia during cesarean delivery by administering local anesthetic agents through a catheter placed in the epidural space without penetrating the dura mater. In this study, epidural anesthesia is operationalized by inserting an 18-gauge Tuohy needle at the L3-L4 lumbar interspace, advancing the epidural catheter 4-5 cm into the epidural space, followed by administration of 0.5% isobaric bupivacaine combined with 50 µg fentanyl. Parameters recorded include sensory and motor block onset, mean arterial pressure (MAP), heart rate, and procedure- and surgery-related adverse events. In this study, epidural anesthetic dosing is adjusted for patients with very short stature (height <150 cm), with dose reduction based on published literature (10-20%).
  Arms: Epidural Anesthesia

SUMMARY:
The goal of this clinical trial is to compare the onset of sensory block between epidural anesthesia and dural puncture epidural (DPE) in patients undergoing elective cesarean delivery. The study also aims to evaluate hemodynamic stability and procedure-related side effects associated with both techniques.

The main questions it aims to answer are:

1. What is the difference in the onset of sensory block between epidural anesthesia and dural puncture epidural (DPE) in patients undergoing cesarean section?
2. Are there differences in hemodynamic stability between epidural anesthesia and DPE during surgery?
3. What procedure-related side effects occur with each anesthetic technique?

Researchers will compare epidural anesthesia with dural puncture epidural (DPE) to determine which technique achieves a faster and more effective sensory block while maintaining maternal hemodynamic stability.

Participants will:

1. Be randomly assigned to receive either epidural anesthesia or DPE anesthesia
2. Undergo elective cesarean delivery under regional anesthesia
3. Have sensory block onset, hemodynamic parameters, and adverse events monitored and recorded intraoperatively

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women scheduled to undergo cesarean delivery
* American Society of Anesthesiologists (ASA) physical status II-III
* Willing to participate in the study by providing written informed consent

Exclusion Criteria:

* Patients with absolute contraindications to neuraxial anesthesia
* Patients with known allergy or history of allergy to medications used in the study
* Patients with psychiatric disorders or who are uncooperative
* Patients with accidental dural puncture

Dropout Criteria:

* Patients who require conversion to general anesthesia during the procedure
* Patients who experience major intraoperative complications (massive hemorrhage, shock, or cardiac arrest)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Time (minutes) to achieve bilateral T6 sensory block | From an anesthetic injection to the achievement of sensory and motor block during surgery (intraoperative period).
  Sensory block onset is defined as the time from anesthetic injection until the achievement of sensory block at the T6 dermatome on both the left and right sides. The measurement is recorded in minutes using a stopwatch.
Time (minutes) to achieve Bromage grade 3 motor block | From an anesthetic injection to the achievement of sensory and motor block during surgery (intraoperative period)
  Motor block onset is defined as the time from anesthetic injection until the achievement of Bromage grade 3 motor block (inability to raise the straight leg). The measurement is recorded in minutes using a stopwatch.

SECONDARY OUTCOMES:
Mean Arterial Pressure (MAP) | From baseline (minute 0) to 20 minutes after anesthetic administration during surgery
  Mean arterial pressure (MAP) is defined as the average arterial blood pressure during a single cardiac cycle and is monitored non-invasively using an automated blood pressure monitor. This parameter is recorded at baseline (minute 0) and subsequently measured every 3 minutes during the first 20 minutes following anesthetic administration.
Heart Rate (HR) | From baseline (minute 0) to 20 minutes after anesthetic administration during surgery
  Heart rate is defined as the number of heartbeats per minute and is measured automatically via standard patient monitoring. Heart rate is recorded at baseline (minute 0) and subsequently measured every 3 minutes during the first 20 minutes following anesthetic administration.
Number of participants with Post-dural Puncture Headache (PDPH) | Within 72 hours after neuraxial anesthesia
  Post-dural puncture headache (PDPH) is assessed as part of the side effect evaluation. PDPH is defined as a postural headache that worsens when the patient is sitting or standing and improves in the supine position, occurring within 48-72 hours after dural penetration. PDPH is evaluated as a secondary outcome as a potential complication following neuraxial anesthesia, including epidural and dural puncture epidural (DPE) techniques.
Number of participants with nausea and/or vomiting | During anesthetic administration and surgery
  Nausea and vomiting are assessed as part of the side effect evaluation. These outcomes are defined as subjective complaints of nausea and/or observed episodes of vomiting occurring during anesthetic administration and throughout the cesarean delivery procedure. Events are assessed through direct observation and patient self-reporting.
APGAR Score | At 1 and 5 minutes after birth
  APGAR Score is assessed as part of the side effect evaluation. Neonatal outcome is assessed using the Apgar score at 1 and 5 minutes after birth. The Apgar score evaluates five parameters: skin color, heart rate, reflex irritability, muscle tone, and respiration, with a total score ranging from 0 to 10. Apgar scores are recorded by trained healthcare personnel and used as an indicator of immediate neonatal clinical condition.
Number of participants with hypotension | From anesthetic administration until the end of surgery
  Hypotension is assessed as part of the side effect evaluation and defined as a decrease in blood pressure of ≥20% from baseline or a mean arterial pressure (MAP) <65 mmHg following neuraxial anesthesia.

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - Dr. Sardjito General Hospital, Sleman, DI Yogyakarta
  - Persahabatan General Hospital, Jakarta, DKI Jakarta

IPD SHARING:
Plan to Share IPD: Undecided